CLINICAL TRIAL: NCT05482204
Title: Do Sustainability Labels Lead to More Sustainable and Healthier Food Choices?
Acronym: Climate Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Time-sharing Experiments for the Social Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00018722
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Food Selection; Attitude
MeSH Terms: conditions — Food Preferences; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (QR) label (No Intervention): QR label on all menu items
- Low Climate Impact Label (Experimental): 'Low Climate Impact' label on all chicken, fish and vegetarian menu items
  Interventions: Other: Low Climate Impact label
- High climate Impact Label (Experimental): 'High Climate Impact' label on all beef menu items
  Interventions: Other: High Climate Impact label

INTERVENTIONS:
Other: Low Climate Impact label — Menu labels indicating low climate impact on chicken, fish, and vegetarian food items on a simulated online fast food menu.
  Arms: Low Climate Impact Label
Other: High Climate Impact label — Menu labels indicating high climate impact on beef food items on a simulated online fast food menu.
  Arms: High climate Impact Label

SUMMARY:
This study tests the effect of two climate change menu labels, one indicating 'low climate impact' and the other indicating 'high climate impact' on ordering choices and perceptions of healthfulness of food ordered in an online randomized experiment.

DETAILED DESCRIPTION:
The objective of this study is to examine how climate impact menu labels influence US adults' ordering and perceptions via an online randomized experiment. Participants were randomized to view one of 3 fast food menus online and then choose an item that they would like to order. One menu 'control' had QR code labels, the second had "low climate impact" labels on items with lower greenhouse gas emissions (vegetarian, chicken or fish items), the third had "high climate impact" labels on beef items. After the ordering task participants answered questions about what label they saw on the menu, how healthy they thought the item they ordered was, and how much the label discouraged them from eating high climate impact items.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Member of the National Opinion Research Center (NORC) Amerispeak Panel

Exclusion Criteria:

* <18 years of age
* completed the survey in < 1/3 of the median duration
* skipped or refused more than 50% of the survey questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5055 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Sustainable vs. unsustainable selection from the menu | 1 minute
  The primary outcome is a binary indicator of whether or not the participant selected during the ordering task was a sustainable (chicken, fish, or vegetarian) menu item (1) vs. an unsustainable (beef) menu item (0).
  Before viewing the fast food menu, participants were asked to imagine they are at a restaurant and about to order dinner. They were asked to select one item they want to order for themselves. Participants could select one item to order before moving on.

SECONDARY OUTCOMES:
Perceptions of healthfulness | < 1 minute
  Perceptions of how healthy the meal ordered was (on a scale of 1=very unhealthy to 7=very healthy)
Perceived Message Effectiveness (PME) | <1 minute
  This outcomes used 1 item from the 3 item UNC-PME scale to measure how much the assigned label discouraged the participant from wanting to consume items with a high impact on climate change. Responses are measured on a 5-point Likert scale from 1=Strongly disagree to 5= strongly agree. The exact question text is: "How much do you agree or disagree with the following statement? Information on the menu discouraged me from wanting to consume menu items with a high impact on climate change."
Nutrition Profile Index of ordered item | < 1 minute
  The Nutrition Profile Index score (0-100) of the ordered item

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Wolfson, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
After 1 year de-identified data will be made available in partnership with the Open Science Foundation.
Supporting Information: Study Protocol
Time Frame: 1 year after study completion.

REFERENCES:
- [Derived] Wolfson JA, Musicus AA, Leung CW, Gearhardt AN, Falbe J. Effect of Climate Change Impact Menu Labels on Fast Food Ordering Choices Among US Adults: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2248320. doi: 10.1001/jamanetworkopen.2022.48320. PMID 36574248